CLINICAL TRIAL: NCT05661279
Title: Ultrasound Guided Rhomboid Intercostal Block Versus Serratus Anterior Plane Block for Analgesia After Thoracodorsal Artery Perforator Flap Following Partial Mastectomy
Brief Title: Rhomboid Intercostal Block Versus Serratus Anterior Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba M Fathi, prof/Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: zu-IRB # 10060
Record Dates: First submitted 2022-12-01; First posted 2022-12-22 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain
Keywords: rhomboid intercostal block -serratus anterior plane block - thoracodorsal artery perforator flap
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C: (Active Comparator): control group who will be given general anesthesia only
  Interventions: Procedure: general anesthesia
- Group R: (Active Comparator): Rhomboid intercostal block then general anesthesia
  Interventions: Procedure: general anesthesia; Procedure: general anesthesia plus Rhomboid intercostal block
- group S (Active Comparator): Serratus anterior plane block then general anesthesia
  Interventions: Procedure: general anesthesia; Procedure: Serratus anterior plane block

INTERVENTIONS:
Procedure: general anesthesia — general anesthesia
Procedure: general anesthesia plus Rhomboid intercostal block — the patients will be positioned in lateral decubitus with moving the scapula laterally by abducting the ipsilateral arm across the chest. under complete aseptic situations A high-frequency (6-12 MHz) linear US probe will be put medial to the medial border of the scapula in an oblique sagittal plane with the orientation marker directed cranially.at the T6-7 level, the tissue plain between the rhomboid major and intercostal muscles is identified, and a single injection of 25mL of bupivacaine (0.25%) will be administered via 18-gauge Tuohy advanced in plane from a superomedial to an inferolateral direction, followed by general anesthesia
  Arms: Group R:
Procedure: Serratus anterior plane block — The patient will be positioned supine with his arm abducts at 90°. the US high frequency (6-12 MHz) linear probe of sonosite M turbo ultrasonography (FUJIFIM sonosite, Inc., Bothell, WA, USA) will be put in sagittal plane at the midaxillary line. identification of the fascial plane between the serratus anterior muscle and external intercostal muscles will be performed between the fourth and fifth ribs in the midaxillary area . At this point the18-gauge Tuohy needle will be advanced in plane with injection of 25mL of 0.25 %, bupivacaine. followed by general anesthesia
  Arms: group S

SUMMARY:
evaluate and compare the impact of ultrasound guided rhomboid intercostal block versus serratus anterior plane block for analgesia after thoracodorsal artery perforator flap following partial mastectomy

DETAILED DESCRIPTION:
* To assess and compare quality of post- operative analgesia in each group.
* Time of performance of block in both groups.
* To assess and compare post-operative hemodynamics as well as anticipated adverse effects including nausea, vomiting, itching, hemorrhage, bradycardia, hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 21 to 60 years
* Undergoing pedicled thoracodorsal artery perforator flap following breast conserving surgery -General anesthesia
* Informed consents
* ASA I & II
* Body mass index 25-30 kg/m2.

Exclusion Criteria:

* patients on anti-platelet, anticoagulant or B blocker drugs
* Patients with acute decompensated heart failure, hypertension, heart block, coronary disease, Asthma, bleeding disorders, compromised renal or hepatic function
* history of allergy to local anesthesia or opioid analgesia,
* pregnancy.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-10-02 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
tramadol consumption | at 24 hours postoperative
  The amount of tramadol consumption

SECONDARY OUTCOMES:
Time of performance of block | time from positioning of ultrasound porbe till the end of block procedure.
  Time needed to performance the block
Time to first dose of rescue analgesia | during the first 24 hours postoperatively
  the first time that the patients need analgesia when VAS ≥ 3
Anticipated side effect | at 24 hous post operative
  nausea, vomiting, local anesthesia toxicity, needle injury
Post operative patient's satisfaction | at 24 hours post operative
  Post operative patient's satisfaction using 3 point scale (1= satisfied ,2=neutral, 3=not satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Fathi, Principal Investigator — faculty of human medicine ,zagazig university
Locations (1):
- Heba M Fathi, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No